CLINICAL TRIAL: NCT04652440
Title: Phase II Study of Ablation Combined With PD-1 Antibody in Patients With Hepatocellular Carcinoma
Brief Title: Ablation Combined With PD-1 in HCC: Phase II Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Min-Shan, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-197-01
Record Dates: First submitted 2020-10-27; First posted 2020-12-03 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Radiofrequency ablation; PD-1 Inhibitor; Hepatocellular Carcinoma; Microwave ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — spartalizumab; tislelizumab

STUDY DESIGN:
Intervention Model Description: Evaluate the safety and tolerability of radiofrequency ablation combined with PD-1 monoclonal antibody in the treatment of patients with hepatocellular carcinoma.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiofrequency or microwave ablation combined with PD-1 monoclonal antibody (Experimental): Patients who meet the inclusion criteria will receive 1 cycle of PD-1 antibody on the day before ablation, then 3 cycles of PD-1 antibody after primary radiofrequency or microwave ablation, on a schedule of per 3 weeks, then be followed until disease relapse or death.
  Interventions: Drug: PD-1 monoclonal antibody; Procedure: Radiofequencey or microwave ablation

INTERVENTIONS:
Drug: PD-1 monoclonal antibody — The enrolled patients received intravenous injections of PD-1 monoclonal antibody (Tislelizumab 200mg) on the 1 day before radiofrequency or microwave ablation treatment, and 21(±7) days, 42(+7) and 63(+7) after ablation.
  Other Names: Tislelizumab
Procedure: Radiofequencey or microwave ablation — The enrolled patients received primary radiofrequency or microwave ablation on the day after the first dose of PD-1 antibody treatment.
  Other Names: ablation

SUMMARY:
This is a Phase 2, single arm, single center study designed to evaluate the safety and tolerability of radiofrequency or microwave ablation combined with PD-1 monoclonal antibody in patients with hepatocellular carcinoma(HCC), with the secondary study objective to preliminarily evaluate the efficacy of radiofrequency or microwave ablation combined with PD-1 monoclonal antibody in patients with HCC and the exploratory study objective to evaluate the effect of ablation combined with PD-1 monoclonal antibody on immune function and hepatitis virus infection status in patients with HCC. This study will be divided into two stages, and the first stage is to enroll 6 patients for dose-limited toxicity (DLT) observation. If DLT appeared in < 2 patients, the second stage was entered and the other 24 patients were further enrolled.

DETAILED DESCRIPTION:
The enrolled patients received intravenous injection of PD-1 monoclonal antibody (tirelizumab 200mg) on the day before ablation and the 21 (± 7) days, the 42 (+ 7) days and the 63 (+ 7) days after ablation, respectively (a total of 4 times). Liver tumor biopsy was performed during ablation, tissue samples will be stored for pathological examination and test of PD-L1 expression.

Liver enhanced MRI or CT and contrast-enhanced ultrasound were reviewed within 4 ~ 6 weeks after the first ablation treatment to evaluate the complete response rate of the tumor after treatment. Patients suspected of local incomplete ablation in either of the two examinations could receive a salvage ablation for once within 12 weeks of the first ablation, but no extra dose of PD-1 antibody would be given. Patients with residual viable tumor after re-ablation were defined as treatment failure.

The first six patients (stage I) underwent detailed physical examination on the 2nd, 7th, 14th and 21st days after receiving the first dose of study drug, and 30 days after the 2nd and 4th doses of study drugs. Blood tests and urine routine were performed on the 2nd day after treatment, as well as ECG examination. In the second stage, the patients underwent examinations on the second and 21st days after the dose of study drug, and on the 30 days after the last dose of study drug (the above examination can be carried out within ± 7 days). If there are clinically significant study related adverse events (including abnormal test results) in patients in stage I, necessary reexamination and visit would be added in patients in stage II.

Radiological evaluation arrangement: liver enhanced MRI or CT and contrast-enhanced ultrasound were performed within 4 ~ 6 weeks after the first ablation. The second imaging examination would be completed within 4 ~ 6 weeks after the end of the study treatment, and then examined according to the following schedule: CT / MRI was repeated every 3 months within the first year, then every 4 months within the next year, and every 6 months after 2 years. The investigators will evaluate the adverse events during the follow-up. After the patients have radiologically confirmed recurrence and/or metastasis, they will be treated according to the guideline without limitation. The information of all anti-cancer treatments they received need to be collected.

Follow-up by phone will be conducted at least every 6 months until death to find out the patient's survival data, as well as their physical condition and information about other anticancer treatment received.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who voluntarily participate in the study and sign the informed consent form
2. 18 ~ 75 years old, both men and women
3. Clinical diagnosis of hepatocellular carcinoma, conforming to the indications of radiofrequency or microwave ablation
4. Child-Pugh score ≤6 (Child-Pugh score A)
5. Barcelona Clinic Liver Cancer (BCLC) Stage A or B
6. Number of tumors ≤ 2; 2 cm<maximum diameter≤ 5 cm
7. No distant metastasis or lymph node metastasis (defined as lymph node maximum transverse diameter ≥ 15 mm)
8. ECOG score 0 or 1
9. No history of drug allergy;
10. The function of vital organs meets the following requirements (no blood component, cell growth factor and other corrective treatment drugs are allowed to be used 14 days before enrollment) 1）Absolute neutrophil count≥1.5×109/L; 2）Platelets≥80×109/L; 3）Hemoglobin≥90 g/L; 4）Serum albumin≥30 g/L; 5）Thyroid stimulating hormone (TSH) ≤1×ULN (if abnormal, FT3 and FT4 should also be investigated, and patients whose FT3 and FT4 levels are normal can be enrolled); 6) Bilirubin≤1.5×ULN (within 7 days prior to the first dose); 7) ALT and AST≤3×ULN (within 7 days prior to the first dose); 8) No prolongation of PT by more than 3 seconds above the ULN; 9)Serum creatinine≤1.5×ULN;
11. Female patients who are not surgically sterilized or of reproductive age need to use contraceptive measures (such as intrauterine device, contraceptives or condoms) during the study treatment period and within 3 months after the end of the study treatment period; female patients of childbearing potential who are not surgically sterilized must have a negative serum or urine HCG test within 72 hours before enrollment; and must be non-lactating; male patients with partners of childbearing potential should take an effective method of contraception during the trial and within 3 months after treatment.

Exclusion Criteria:

1. Patients unsuitable for percutaneous radiofrequency or microwave ablation for any reason
2. Any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism; vitiligo; patients with complete remission of asthma in childhood but requiring no intervention after adulthood can be included; patients with asthma requiring medical intervention with bronchodilators can not be included)
3. Patients who need to use immunosuppressive agents or require systemic hormone therapy to achieve the purpose of immunosuppression (dose > 10 mg/day prednisone or other effective hormones) and are still using them within 2 weeks before enrollment
4. Prior systemic anticancer therapy
5. Received or intended to receive other anticancer therapy (vascular intervention, etc.) other than surgical resection or ablative therapy
6. Known history of central nervous system metastasis or hepatic encephalopathy
7. Tumor necrosis cannot be confirmed by reexamination of imaging after local ablation
8. Clinically symptomatic ascites requiring puncture and drainage or those who have received ascites drainage in the past 3 months, except those with only a small amount of ascites shown by imaging but not accompanied by clinical symptoms
9. Hypertension not well controlled by antihypertensive medication (systolic blood pressure≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg)
10. Uncontrolled cardiac clinical symptoms or diseases, such as: (1) heart failure above NYHA2; (2) unstable angina; (3) myocardial infarction within 1 year; (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention; (5)QTc > 450 ms (male); QTc > 470 ms (female)
11. Abnormal coagulation function (INR > 2.0, PT > 16s), bleeding tendency or receiving thrombolytic or anticoagulant therapy. Prophylactic use of low-dose aspirin and low-molecular-weight heparin is allowed
12. Patients with clinically significant bleeding symptoms or bleeding tendency within 3 months before randomization, such as hemoptysis more than 2.5ml per day, gastrointestinal bleeding, esophageal and gastric varices at risk of bleeding, hemorrhagic gastric ulcer, vasculitis, etc. If the stool occult blood is positive at baseline, reexamination must be performed. if it is still positive after reexamination, gastroscopy is required. If gastroscopy suggests severe esophageal and gastric varices, patients can't be enrolled (except for those who receive gastroscopy to rule out such conditions within 3 months before enrollment)
13. Arterial/venous thrombotic events occurred within 6 months before enrollment, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism
14. Known hereditary or acquired bleeding and thrombophilia (such as hemophilia, coagulation dysfunction, thrombocytopenia, etc.)
15. Urine routine test showed urine protein≥+ + and 24-hour urine protein > 1.0 g is confirmed
16. Patients who previously received radiotherapy, chemotherapy and hormone therapy for anti-cancer
17. Patients with active infection or fever of unknown origin 7 days before the first dose, T≥38℃, or baseline white blood cell count > 15×109/L
18. Patients with congenital or acquired immunodeficiency (such as HIV infection)
19. Untreated active hepatitis virus infection with HBV DNA > 2000 IU/m (l or 104 copies/ml), HCV RNA > 103 copies/ml
20. Patients with other malignant tumors (except cured cutaneous basal cell carcinoma and carcinoma in situ of cervix) within 3 years previously or simultaneously
21. Patients who have other factors that may affect the study results or cause the study to be halted, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring concomitant treatment, severe laboratory abnormalities, with family or social factors that may affect the safety and compliance of patients as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Measure Safety | from the start of PD-1 monoclonal antibody therapy to 90 days after treatment
  Treatment-related adverse events (TRAEs) and serious adverse events (SAEs) occurring from the start of PD-1 monoclonal antibody therapy to 90 days after treatment were observed and judged according to CTCAE 5.0 criteria.
Measure Tolerability | from the start of PD-1 monoclonal antibody therapy to 90 days after treatment
  Measured as the rate of patients able to complete treatment as planned in the study.

SECONDARY OUTCOMES:
Complete Response (CR1) | Two years
  Complete response rate of single ablation combined with PD-1 monoclonal antibody in patients with hepatocellular carcinoma
Treatment Failure Rate (TFR) | Two years
  Rate of treatment failure (rate of patients with lesions residue after first ablation and tumor survival after re-ablation)
Local Recurrence Rate (LRR) and Distant Metastasis Rate (DMR) | Two years
  1- and 2-year local recurrence rate (LRR) and distant metastasis rate (DMR) after ablation
1- and 2-year disease-free survival (DFS) and overall survival (OS) rates | Two years
  The percentage of patients who were without disease or still alive at the 1- and 2-year time point since the first cycle of treatment. The end point of observation is death due to tumor.
Median Disease-free survival (mDFS) | Two years
  median disease-free survival of patients after ablation

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Will share the data on https://www.researchdata.org.cn/default.aspx.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: 1 year after the study complete.
URL: https://www.researchdata.org.cn/default.aspx